CLINICAL TRIAL: NCT05942469
Title: Fostering Optimal Regulation of Emotion for Prevention of Secondary Trauma (FOREST): Implementation and Evaluation of a Burnout Prevention Program for Staff in Gun Violence Prevention Programs
Brief Title: Fostering Optimal Regulation of Emotion for Prevention of Secondary Trauma (FOREST)
Acronym: FOREST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Judith Moskowitz, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00219630
Record Dates: First submitted 2023-06-26; First posted 2023-07-12 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Burnout; Burnout, Professional; Positive Affect; Depression; Anxiety; Compassion Fatigue; Job Stress
Keywords: Burnout; Anxiety; Depression; Positive Emotion; Coping; Job Stress
MeSH Terms: conditions — Burnout, Psychological; Burnout, Professional; Depression; Anxiety Disorders; Compassion Fatigue; Occupational Stress | interventions — Forests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOREST + Assessments (Experimental): UCAN staff will participate in Monthly Skill Sessions and complete FOREST content modules in the Learning Management System (LMS). Staff will also be invited to complete annual assessments for primary and secondary outcome measures, as well as annual interviews and focus groups to gather feedback on progress, implementation, and content.
  Interventions: Behavioral: FOREST

INTERVENTIONS:
Behavioral: FOREST — The skill sessions will include didactic content defining the skill, rationale for including the skill in FOREST, and research demonstrating that practice of the skill increases positive emotion. In addition, the group will practice the skill together and will discuss ways to practice the skill at work as well as outside of work. Throughout the month, PEAs will implement the FOREST skill of the month in other existing meetings, check-ins, and team outings.
  Concurrently, a module in UCAN's learning management system (LMS) will become available. The LMS modules will contain skill-related content similar to what is taught in the skill sessions, including a thorough definition of the skill, examples of ways to utilize the skill, a review or summary of the skill, and several knowledge questions to check for comprehension. The LMS content may include text, audio, images, and video components.

SUMMARY:
FOREST is a positive emotion skills program designed to target mental health and coping needs for frontline violence prevention workers at UCAN. Ten skills are taught over a period of nine months during existing meetings and wellness activities, as well as in online modules in UCAN's Learning Management System (LMS). Through infusing the FOREST skills throughout UCAN, we hope to inspire organizational culture change that will emphasize the importance of wellbeing and enhance resilience, therefore reducing burnout and turnover.

DETAILED DESCRIPTION:
All frontline UCAN staff will receive the FOREST program. Each month for 9 months there will be a focus on one to two positive emotion skills. The skill(s) of the month will be taught to the staff during existing one-hour wellness meetings/activities, and will be co-facilitated by Positive Emotion Ambassadors (PEAs; UCAN Staff members nominated to infuse the skills into UCAN culture) and Northwestern University.

The skill sessions will include didactic content defining the skill and explaining the rationale for inclusion, as well as examples of existing research demonstrating the skills benefits. During the session the group will practice the skill together and discuss ways to use the skill in both work and personal situations. Throughout the month, PEAs will implement the FOREST skill of the month in other existing meetings, check-ins, and team outings

The monthly sessions will be observed by a member of the Implementation Resource Team (IRT) who will use a checklist to track that all core pieces of the skill training were delivered. Once a month, the IRT will meet with the PEAs for additional training and support. These sessions will be audio recorded for qualitative data on facilitators and barriers to the skill.

Each month a module in UCAN's learning management system (LMS) that covers that month's skill(s) will also become available. The LMS modules will contain skill-related content similar to what is taught in the skill sessions, including a thorough definition of the skill, examples of ways to utilize the skill, a review or summary of the skill, and several knowledge questions to check for comprehension. The LMS content may include text, audio, images, and video components. All UCAN frontline CVI staff will be required to complete the LMS FOREST skill module of the month. Percentage of staff completing each LMS training will be tracked.

Annual assessments to assess primary and secondary outcomes will be administered via REDCap. Annual interviews and focus groups will ask for feedback on implementation and content.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Currently employed by UCAN
* Has internet access
* Speaks and reads English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Decrease in burnout measured by the Maslach Burnout Inventory (MBI). | 12 months
  The MBI evaluates burnout severity based on three aspects: emotional exhaustion, depersonalization, and lack of personal accomplishment, with higher scores on the emotional exhaustion and depersonalization subscales, and lower scores on the personal accomplishments subscale, indicating increased levels of burnout. Responses on the scale range from "never" to "every day."
Increase in positive affect measured by PROMIS Short Form v1.0- Positive Affect 15a. | 12 months
  PROMIS Positive Affect assesses momentary positive or rewarding affective experiences, such as feelings and mood associated with pleasure, joy, elation, contentment, pride, affection, happiness, engagement, and excitement. Responses options range from "Not at all" to "Very much" with higher scores indicate higher levels of positive affect.
Decrease in depression measured by PROMIS Short Form v1.0- Depression 4a. | 12 months
  PROMIS Depression Bank assesses self-reported negative mood (sadness, guilt), views of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). Response options range from "Never" to "Always" with higher scores indicate higher levels of depression.
Decrease in anxiety measured by PROMIS Short Form v1.0- Anxiety 4a. | 12 months
  PROMIS Anxiety Bank assesses self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). Response options range from "Never" to "Always" with higher scores indicate higher levels of anxiety.
Measure of trauma exposure using the Lifetime Events Checklist (LEC). | 12 months
  The LEC measures trauma exposure, including the ability to differentiate direct experience vs work-related or other secondary exposure through a series of questions about stressful events, with responses including "happened to me," "witnessed it," "learned about it," "not sure," and "doesn't apply," followed up by a question asking if the experience happened as part of one's job. There is no formal scoring protocol or interpretation per se, other than identifying whether a person has experienced one or more of the events listed.
Measure of PTSD symptoms using the the PTSD Checklist for DSM-5 (PCL-5). | 12 months
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Responses range from "not at all" to "extremely," with higher scores indicating higher occurrence of PTSD symptoms.
Increase in meaning and purpose measured by PROMIS Short Form v1.0- Meaning and Purpose 4a. | 12 months
  PROMIS Meaning and Purpose Bank assesses one's sense of life having purpose and that there are good reasons for living. Higher scores indicate hopefulness, optimism, goal-directedness, and feelings that one's life is worthy.
Improvement in professional quality of life/well-being measured by Eudaimonic Workplace Well-being Scale (EWWS). | 12 months
  EWWS measures workplace well-being on both interpersonal and intrapersonal dimensions through a series of eight statements where respondents indicate how strongly they relate to those statements. Values range from "strongly disagree" to "strongly agree," with higher scores reflecting higher workplace well-being/quality of life.

SECONDARY OUTCOMES:
Decrease in staff turnover. | 12 months
  Measured by number of UCAN staff who have left their job after <1 year of employment based on employee records
Increase in staff retention | 12 months
  Measured by number of staff who have stayed employed for >1 year based on employee records
Increase in staff promotion | 12 months
  Measured by number of staff who have been promoted into a new role based on employee records
Decrease in use of sick days | 12 months
  Measured by average number of sick days used per staff member based on employee records

CONTACTS AND LOCATIONS:
Overall Officials: Judith Moskowitz, PhD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States